CLINICAL TRIAL: NCT03742440
Title: GrafixPL PRIME Evaluation Case Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Osiris Therapeutics (Industry)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022018-035
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Results first posted 2020-07-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GrafixPL PRIME (Other): Open-label case series to evaluate GrafixPL PRIME. All subjects receive the product.
  Interventions: Biological: GrafixPL PRIME

INTERVENTIONS:
Biological: GrafixPL PRIME — GrafixPL PRIME

SUMMARY:
The investigators plan to evaluate healing in a cohort of patients with chronic wounds (n=40) that receive optimal treatment including serial wound debridement and off-loading with total contact casts or a boot and GrafixPL PRIME. In addition, the investigators will collect data on other potential confounding factors that could affect healing such as medications, tobacco, nutrition, comorbidities, diabetes control, infection, perfusion, and activity. Wound healing, including wound size and adverse events will be evaluated. The objective of this study is to understand the use of this product to evaluate wound healing in 40 patients.

DETAILED DESCRIPTION:
Screening and Enrollment:

* Review and sign the Informed Consent and HIPAA Authorization
* Review the inclusion and exclusion criteria

If the subject qualifies for the study, they will participate in the following procedures (weekly visits, +/-4 days):

Visit 0:

* Demographics (such as age, gender, race or ethnicity)
* Medical/Surgical and Social History, Current Antibiotics.
* Laboratory Results
* Vascular - ABI
* Neurological evaluation - Monofilament and VPT
* Vitals - Sitting blood pressure and Pulse rate, Height/Weight, and BMI
* Wound debridement
* eKare - Wound imaging measurement
* Application of GrafixPL PRIME
* Current Antibiotics
* Offloading
* Adverse Events
* Source documentation

Visits 1 - 11:

* Wound debridement
* eKare - Wound imaging measurement
* Application of GrafixPL PRIME
* Current Antibiotics
* Offloading
* Adverse Events
* Source documentation

Visit 12/End of Study (EOS) Visit:

* Wound debridement
* eKare - Wound imaging measurement
* Current Antibiotics
* Offloading
* Adverse Events
* Source documentation (End of Study will occur on the date the subject is healed)

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 18-90 years of age
* Chronic foot ulceration below the ankle - persistent for 30 days or longer
* Ankle Brachial Index (ABI) >0.5 (Bedside ABI is acceptable for screening purposes as the formal imaging ABI may not be resulted prior to surgery)

Exclusion Criteria:

* Unable to provide informed consent
* <18 or >90 years of age
* History of poor compliance with follow-up visits
* Gangrene
* Untreated Osteomyelitis
* Widespread malignancy
* Active alcohol or substance abuse such as cocaine, heroin, or methamphetamines
* Currently Pregnant or planning pregnancy during the course of intended participation in the study
* Is nursing or actively lactating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GrafixPL PRIME
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: feet
Arm/Group | GrafixPL PRIME
Number analyzed (Participants) | 40
Number analyzed (feet) | 40
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age of All Participants | 61 (36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 25
  Race: African American | 7
  Race: Hispanic | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Closure of the Index Ulcer
Description: Complete closure of the index ulcer, defined as 100% re-epithelialization as determined by the Investigator by week 12 or the End of Treatment Visit.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GrafixPL PRIME
Number analyzed (Participants) | 40
Participants | 19

2. Secondary Outcome: Time to Closure
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GrafixPL PRIME
Number analyzed (Participants) | 40
days | 40.0 (20.1)

3. Secondary Outcome: Total Adverse Events
Description: There was no control arm in this study - everyone enrolled received treatment. Analysis of these data was separated into two groups - "closed wounds" and "not closed wounds." Wounds that closed achieved full epithelialization within the 12 week study time frame. Wounds that did not close did not achieve full epithelialization by the end of study visit.
Time Frame: 12 weeks
Population: There was no control arm in this study. Analysis of these data was separated into two groups - "closed wounds" and "not closed wounds." Wounds that closed achieved full epithelialization within the 12 week study time frame. Wounds that did not close did not achieve full epithelialization by the end of study visit.
Measure: Number; unit: number of adverse events
Arm/Group | GrafixPL PRIME
Number analyzed (Participants) | 40
number of adverse events
  Closed: number analyzed (Participants) | 19
  Closed | 6
  Not closed: number analyzed (Participants) | 21
  Not closed | 17

ADVERSE EVENTS:
Time Frame: 12 weeks of weekly visits
Groups:
- GrafixPL PRIME: Open-label case series to evaluate GrafixPL PRIME. All subjects received the product.
  GrafixPL PRIME: GrafixPL PRIME
Arm/Group | GrafixPL PRIME
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GrafixPL PRIME (N=40)
Hospitalized for foot-related issue (Surgical and medical procedures) | 2 (2)
Non-foot related hospitalization (Infections and infestations) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GrafixPL PRIME (N=40)
All adverse events (Infections and infestations) | 23 (23) — Includes all reinfections of the foot, pneumonia, antibiotics for any reason not including foot infection, and cutaneous abscess on non-study limb.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03742440/Prot_ICF_001.pdf